CLINICAL TRIAL: NCT04749290
Title: Comparative Effects of Cow's Milk Based Infant Formula Containing Both OPO and CPP Versus Non-OPO Formula and Breast Feeding on Growth, Stool Consistency and Bone Strength: A Double-blinded, Randomized and Controlled Study
Brief Title: Effects of an Infant Formula on Growth, Safety and Efficacy for Healthy Term Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bunge Loders Croklaan (Industry)
Collaborators: Junlebao Dairy Group Co., Ltd. (Industry); Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 20-SM-09-Bunge-001
Record Dates: First submitted 2021-01-30; First posted 2021-02-11 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Infant Development

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study Formula (Experimental): a Cow's Milk Based Infant Formula Containing Both OPO and CPP for term infants (JunLeBao ZhiZhen)
  Interventions: Other: Study Formula
- Comparator Formula (Active Comparator): Commercially available infant formula without OPO for term infants (JunLeBao LeChun)
  Interventions: Other: Study Formula
- Human Milk Reference Group (No Intervention): Human milk

INTERVENTIONS:
Other: Study Formula — Study infant formula for term infants containing OPO and CPP
  Arms: Comparator Formula; Study Formula

SUMMARY:
The purpose of this study is to evaluate that a Cow's Milk Based Infant Formula A2 Containing Both OPO and CPP for healthy term infants supports age-appropriate growth. In this randomized, controlled trial (RCT), healthy, term, formula-fed (FF) infants will be randomized to one of two infant formulas: a standard, commercially-available infant formula for term infants (CF) or the study formula for term infants (SF) for 16 weeks. A reference group of human milk-fed infants will also be enrolled. The primary objective is to compare the growth, tolerance, stool consistency and bone strength of infants randomized to the study infant formula (SF) versus infants randomized to the standard commercial infant formula (CF).

DETAILED DESCRIPTION:
This study is a randomized, controlled, double-blind, study of healthy term formula fed (FF) infants. FF infants will be randomized to receive either a study infant formula, formulated for healthy term infants or a commercially available infant formula for healthy term infants. Infants will consume the formula for a total of 16-weeks; infant growth, tolerance, stool consistency and bone strength will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* 30 days of age at randomization, inclusive (day of birth is considered day 0)
* Exclusively formula-fed or partially bottle feeding with intake more than 650 ml /day for at least 3 days prior to randomization
* Exclusively breast fed for at least 7 days prior to randomization
* Singleton birth
* Gestational age of 37-42 weeks (36 weeks and six days is considered 36 weeks of gestational age)
* Birth weight of 2500g to 4000g
* Signed informed consent obtained for infant's participation in the study
* Parent or guardian of infant agrees not to enroll infant in another interventional clinical research study while participating in this study

Exclusion Criteria:

* History of underlying metabolic or chronic disease; congenital malformation; or any other condition which, in the opinion of the Investigator, is likely to interfere with: the ability of the infant to ingest food, the normal growth and development of the infant, or the evaluation of the infant
* Evidence of feeding difficulties or formula intolerance, such as vomiting or poor intake, at time of randomization (at investigator discretion)
* Weight at Visit 1 is <95% of birth weight [(weight at Visit 1÷birth weight) x 100 <95%]
* Infant is immunocompromised (according to a doctor's diagnosis of immunodeficiency such as Combined Immunodeficiencies, DiGeorge Syndrome, Wiskott-Aldrich Syndrome, Severe Congenital Neutropenia and Secondary Immunodeficiencies linked to HIV infection, Down Syndrome or others) and children with known head/brain disease/injury such as Microcephaly, Macrocephaly or others
* Participation in another clinical trial
* Known or increased risk of cow's milk allergy and/ or lactose intolerance (i.e. one of the biological parents and or siblings diagnosed with cow's milk allergy, asthma, hay fever, etc.)
* Having a mother suffering from diabetes during pregnancy
* Use of antibiotics at the time of screening, or during the past two weeks

Ages: 14 Days to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Stool characteristics | 1 month to 5 months
  Infant Stool Form Scale to measure stool consistency, amount and color (Bekkali et al, 2009): 4-point scale as watery (A) soft (B) formed (C) or hard (D)

SECONDARY OUTCOMES:
Formula intake and tolerance (24 hour dietary recall) | 2 months to 5 months
  ml /day
Medically-diagnosed adverse events collected throughout the study period | 1 month to 5 months
  frequency
Crying and sleep tracking (24 hours recall) | 2 months to 5 months
  frequency
Gastrointestinal tract discomfort | 1 month to 5 months
  frequency of parents observed and documented GI tract discomfort
Anthropometric parameters on growth | 1month to 5 months
  Achieved body length (CM)
Anthropometric parameters on growth | 1month to 5 months
  Achieved head circumferences (CM)
Anthropometric parameters on growth | 1month to 5 months
  Achieved body weight (kg)
Bone Speed Of Sound | at 1 month and 5 months
  Ultrasound Bone Densitometer (BMD-A3)
Anthropometric parameters on growth | 1month to 5 months
  Rate of gain (%) on achieved head circumferences
Anthropometric parameters on growth | 1month to 5 months
  Rate of gain (%) on achieved body weight
Anthropometric parameters on growth | 1month to 5 months
  Rate of gain (%) on achieved body length

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyang Shen, MD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (2):
- China (2):
  - JiangNan Street Community Health Service Center, WuCheng District, Jinhua
  - QiuBin Street Community Health Service Center, WuCheng District, Jinhua

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sheng XY, Mi W, Yuan QB, Liu BY, Carnielli V, Ning YB, Einerhand AWC. An A2 beta-casein infant formula with high sn-2 palmitate and casein phosphopeptides supports adequate growth, improved stool consistency, and bone strength in healthy, term Chinese infants: a randomized, double-blind, controlled clinical trial. Front Nutr. 2024 Aug 14;11:1442584. doi: 10.3389/fnut.2024.1442584. eCollection 2024. PMID 39206307